CLINICAL TRIAL: NCT02218073
Title: A Single-Dose, Open-Label, Randomized, Two-Way Crossover Pharmacokinetic Study to Assess the Relative Bioavailability of Orally Administered JNJ-42756493 Following Intake of a Tablet Versus a Solution and to Assess the Absolute Bioavailability of Orally Administered JNJ-42756493 Following Concomitant Administration of an Intravenous Microdose of the Stable Isotope JNJ-61818549 in Healthy Subjects
Brief Title: Pharmacokinetic Study of JNJ-42756493 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR104998; 42756493EDI1002 (Other: Janssen Research & Development, LLC); 2014-002634-31 (EudraCT Number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42756493; JNJ-61818549; Isotope
MeSH Terms: interventions — erdafitinib; Tablets; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive 10 milligram (mg) JNJ-42756493 tablet orally on Day 1 of Period 1 and 100 microgram (mcg) of JNJ-61818549 as intravenous injection 2 hours after the intake of 10 mg JNJ-42756493 oral solution on Day 1 of Period 2.
  Interventions: Drug: JNJ-42756493 10 mg tablet; Drug: JNJ-42756493 10 mg Oral Solution; Drug: JNJ-61818549
- Treatment Sequence BA (Experimental): Participants will receive 100 mcg of JNJ-61818549 as intravenous injection after the intake of 10 mg JNJ-42756493 oral solution on Day 1 of Period 1 and JNJ-42756493 10 mg tablet orally on Day 1 of Period 2.
  Interventions: Drug: JNJ-42756493 10 mg tablet; Drug: JNJ-42756493 10 mg Oral Solution; Drug: JNJ-61818549

INTERVENTIONS:
Drug: JNJ-42756493 10 mg tablet — Participants will be administered with 10 milligram (mg) JNJ-42756493 tablet orally either on Day 1 of Period 1 or on Day 1 of Period 2.
Drug: JNJ-42756493 10 mg Oral Solution — Participants will be administered with 10 mg JNJ-42756493 oral solution either on Day 1 of Period 1 or on Day 1 of Period 2.
Drug: JNJ-61818549 — Participants will receive 100 mcg of JNJ-61818549 as intravenous injection on Day 1 of Period 2 or Day 1 of Period 1.

SUMMARY:
The purpose of this study is to evaluate the absolute bioavailability (the extent to which a drug or other substance becomes available to the body) of JNJ-42756493 following a single 10 milligram (mg) dose as an oral solution administered in combination with a single intravenous administration of a microdose (100 microgram [mcg]) of JNJ-61818549 and to evaluate the relative bioavailability of 10 mg JNJ-42756493 following an oral solution (reference) and a tablet (test) formulation in a crossover (method used to switch subjects from one study group to another in a clinical trial) design in healthy participants.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all people know the identity of the intervention), 2-way crossover, single-dose, and single-center, Phase 1 study of oral JNJ-42756493 in healthy participants. The duration of the study is approximately 36-63 days: 2-20 days Screening, two 7 days open-label treatment periods, 12-14 days washout and 12-14-day follow-up (Day 13-15 of period 2). All participants will be randomly assigned to 1 of 2 treatment sequences. In Treatment Sequence AB: JNJ-42756493 10 mg tablet formulation will be administered on Day 1 of Period 1 and 100 mcg JNJ-61818549 will be administered intravenously 2 hours after the intake of 10 mg JNJ-42756493 oral solution on Day 1 of Period 2. In Treatment Sequence BA: 100 mcg JNJ-61818549 will be administered intravenously after the intake of 10 mg JNJ-42756493 oral solution on Day 1 of Period 1 and 10 mg JNJ-42756493 tablet formulation will be administered on Day 1 of Period 2. A minimum 12 days washout is required between treatment periods. Participants will primarily be analyzed for pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Received a thorough explanation of the optional pharmacogenomic research component of the study and was offered an opportunity to participate by signing the separate pharmacogenomic informed consent document
* If a woman, must be postmenopausal (no spontaneous menses for at least 2 years), or surgically sterile
* If a woman, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening
* Body mass index (BMI) (weight kilogram [kg]/ height square meter[m^2] between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kg
* Non-smoker for at least 6 months before entering the study

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, metabolic bone disease (other than osteoporosis), infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening and predose on Day -2 (urinalysis only) and on Day -1 of both treatment Period as deemed appropriate by the investigator. Retesting of abnormal lab values that may lead to exclusion will be allowed once
* Clinically significant abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) at screening and Day -1 of both treatment Periods as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability: Maximum Plasma Concentration (Cmax) | Day 1 (pre-dose); 15, 30 and 60 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, 72, 96, 120 and 144 hours post-dose
  The Cmax is the maximum observed plasma concentration of JNJ-42756493.
Absolute Bioavailability | Day 1 (pre-dose); 15, 30 and 60 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, 72, 96, 120 and 144 hours post-dose
  Absolute bioavailability will be measured by Area under concentration time-curve (AUC [0-24]), AUC (0-last) and AUC (0-infinity).
Relative Bioavailability: Area under concententration time-curve (AUC) | Day 1 (pre-dose); 15, 30 and 60 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, 72, 96, 120 and 144 hours post-dose
  Relative bioavailability will be measured by AUC (0-24), AUC (0-last) and AUC (0-infinity).

SECONDARY OUTCOMES:
Time to Reach Maximum Concentration (tmax) | Day 1 (pre-dose); 15, 30 and 60 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, 72, 96, 120 and 144 hours post-dose
  The tmax is time to reach the maximum observed plasma concentration.
Elimination Half-Life (t1/2) | Day 1 (pre-dose); 15, 30 and 60 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, 72, 96, 120 and 144 hours post-dose
  Terminal phase elimination half-life is the time measured for the serum concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium